CLINICAL TRIAL: NCT05844046
Title: Sequential or Up-front Triple Treatment With Durvalumab, Tremelimumab and Bevacizumab for Non-resectable Hepatocellular Carcinoma (HCC) Patients (MONTBLANC)
Brief Title: Sequential or Up-front Triple Treatment With Durvalumab, Tremelimumab and Bevacizumab for Non-resectable Hepatocellular Carcinoma (HCC) Patients
Acronym: MONTBLANC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Enrico De Toni (Other)
Responsible Party: Sponsor-Investigator, Enrico De Toni, Prof. Dr. Enrico De Toni, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MONTBLANC; 2022-001201-48 (EudraCT Number)
Record Dates: First submitted 2023-04-11; First posted 2023-05-06 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — durvalumab; tremelimumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Durvalumab (1500 mg q4w) plus tremelimumab (300 mg x 1) followed by addition of bevacizumab (15mg/kg) upon detection of radiological progression or in the absence of objective response after the second staging.
  Interventions: Biological: durvalumab, tremelimumab, bevacizumab
- Arm B (Experimental): Durvalumab plus tremelimumab followed by maintenance treatment with durvalumab and bevacizumab.
  Interventions: Biological: durvalumab, tremelimumab, bevacizumab

INTERVENTIONS:
Biological: durvalumab, tremelimumab, bevacizumab — durvalumab, tremelimumab and bevacizumab will be administered in the respective arms either as up-front triple treatment or as combined treatment with durvalumab and tremelimumab followed by the addition of bevacizumab

SUMMARY:
This is a randomized, open-label, multi-center, international, Phase II study to assess the efficacy and safety of sequential or up-front triple treatment with durvalumab, tremelimumab and bevacizumab for non-resectable hepatocellular carcinoma.

Patients will be randomized in a 1:1 ratio to one of the following arms:

Arm A: initial treatment with durvalumab plus tremelimumab followed by treatment escalation with the addition of bevacizumab upon radiological progression or in the absence of objective response

Arm B: up-front treatment with durvalumab, tremelimumab and bevacizumab

Patients will be stratified according to macrovascular invasion and etiology of liver disease (viral etiologies versus others).

ELIGIBILITY:
KEY INCLUSION CRITERIA

Age ≥18 years at the time of study entry

Confirmed HCC based on histopathological findings from tumor tissues.

Must not have received prior systemic therapy for HCC.

Not eligible for locoregional therapy for unresectable HCC. For patients who progressed after locoregional therapy for HCC, locoregional therapy must have been completed ≥28 days prior to the baseline scan for the current study.

Barcelona Clinic Liver Cancer (BCLC) stage B (that is not eligible for locoregional therapy) or stage C

Child-Pugh Score class A

ECOG performance status of 0 or 1 at enrollment

At least 1 measurable lesion, not previously irradiated, that can be accurately measured at baseline as ≥10 mm in the longest diameter (except lymph nodes, which must have a short axis ≥15 mm) with computerized tomography (CT) or magnetic resonance imaging (MRI), and that is suitable for accurate repeated measurements as per RECIST 1.1 guidelines. A lesion which progressed after previous ablation or TACE could be measurable if it meets these criteria.

Adequate organ and marrow function

KEY EXCLUSION CRITERIA

Previous study drug(s) assignment in the present study.

Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 28 days of the first dose of study drug(s).

Major surgical procedure or significant traumatic injury within 28 days prior to the first dose of study drug(s), abdominal surgery, abdominal interventions, or significant abdominal traumatic injury within 60 days prior to randomization

History of allogeneic organ transplantation (eg, liver transplant).

History of hepatic encephalopathy within past 12 months or requirement for medications to prevent or control encephalopathy

Clinically meaningful ascites

Patients with main portal vein thrombosis (i.e., thrombosis in the main trunk of the portal vein, with or without blood flow) on baseline imaging.

Patient currently exhibits symptomatic or uncontrolled hypertension

Active or prior documented autoimmune or inflammatory disorders, diverticulitis. Patients without active disease in the last 5 years are excluded unless discussed with the Study Physician and considered appropriate for study participation.

Patients co-infected with HBV and HCV, or co-infected with HBV and hepatitis D virus (HDV).

History of another primary malignancy except for the exceptions defined by the study protocol.

Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart).

Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.

History of active primary immunodeficiency.

Receipt of live attenuated vaccine within 30 days prior to the first dose of study drug(s). Note: Patients, if enrolled, should not receive live vaccine while receiving study drug(s) and up to 30 days after the last dose of study drug(s).

Major gastrointestinal bleeding within 4 weeks prior to randomization.

Patients with untreated or incompletely treated varices with bleeding or high-risk for bleeding. Patients must undergo an esophagogastroduodenoscopy (EGD), and all size of varices (small to large) must be assessed and treated per local standard of care prior to enrollment. Patients who have undergone an EGD within 6 months prior to randomization do not need to repeat the procedure. Those who have received banding and/or sclerotherapy and with no bleeding event within the prior 6 months are eligible provided that a re-endoscopy is performed and that varices remained obliterated, minimal or Grade I

Significant vascular disease including aortic aneurysm requiring surgical repair or peripheral arterial thrombosis with 6 months prior to randomization

History of abdominal or tracheoesophageal fistula or gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to randomization.

Evidence of bleeding diathesis or significant coagulopathy

Severe, nonhealing or dehisced wound, active ulcer, or untreated bone fracture

Current or recent (within 10 days of randomization) use of acetylsalicyclic acid (=> 325 mg/day) or treatment with dipyramidole, ticlopidine, clopidogrel, and cilostazol

Current or recent (within 10 days prior to randomization) use of fulldose oral or parenteral anticoagulants or thrombolytic agents for therapeutic purpose. Prophylactic use of low molecularweight heparin is allowed.

Female patients who are pregnant or breastfeeding, or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy or 180 days after the last dose of durvalumab plus tremelimumab combination therapy or bevacizumab therapy

Prior randomization or treatment in a previous durvalumab and/or tremelimumab clinical study regardless of treatment arm assignment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2023-04-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 24 months
  overall response rate

SECONDARY OUTCOMES:
mOS | 24 months
  median overall survival
PFS | 24 months
  Progression-free survival
TTP | 24 months
  Time to progression
ORR-BICR | 24 months
  Objective response rate acc. to BICR

OTHER OUTCOMES:
DOR | 24 months
  Duration of response
DCR | 24 months
  Disease control rate
OS-18m | 18 months
  Proportion of patients alive at 18 months
OS-24m | 24 months
  Proportion of patients alive at 24 months
PFS-E | 24 months
  Progression-free survival from escalation treatment
PFS on next treatment | 24 months
  PFS on next treatment
TTFS | 24 months
  time to failure of strategy
QOL | 24 months
  European Organisation for Research and Treatment of Cancer (EORTC) 30-item core quality of life questionnaire (QLQ-C30)
QOL | 24 months
  EORTC 18-item hepatocellular carcinoma quality of life questionnaire

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Hospital of the University of Munich, Munich
  - Klinikum Rechts der Isar of the Technical University Munich, Munich
  - Würzburg University Hospital, Würzburg

REFERENCES:
- [Background] De Toni EN, Mayerle J, Oehrle B, Seidensticker M, Rimassa L, Philipp A, Roessler D, Khaled NB. Letter: Presence of progression or absence of response? Alternative trial designs for immunotherapy of advanced hepatocellular carcinoma. Aliment Pharmacol Ther. 2024 Jun;59(11):1462-1464. doi: 10.1111/apt.17985. Epub 2024 Apr 21. No abstract available. PMID 38643505